CLINICAL TRIAL: NCT03095417
Title: Decreasing Alzheimer's Disease and Related Dementias After Delirium- Exercise and Cognitive Training
Brief Title: Improving the Recovery and Outcome Every Day After the ICU
Acronym: IMPROVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Babar Khan, MD, MS, Assistant Professor of Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1608126693; R01AG055391 (NIH)
Record Dates: First submitted 2017-03-23; First posted 2017-03-29 (Actual); Results first posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-02

CONDITIONS: Delirium; Alzheimer Disease
Keywords: Delirium; Alzheimer's Disease; Aging; Exercise Therapy; Cognitive Training
MeSH Terms: conditions — Delirium; Alzheimer Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Physical Exercise and Cognitive Training (Experimental): Physical Exercise Intervention: The physical exercise portion of the combined intervention consists of 45 minutes of multi-modal physical exercise focused on seated aerobic and progressive resistance training designed to improve aerobic capacity, muscular strength and endurance consistent with current exercise recommendations. The study team will deliver 3 sessions per week for 3 months.
  Cognitive Intervention: The cognitive portion of the combined intervention consists of a suite of 24 programs called Brain HQ developed by Posit Science Inc., organized into six categories: attention, speed, memory, people skills, intelligence, and navigation. The DDD-ECT trial will use 45-minute sessions of Brain HQ exercises. The modules are designed to improve time-order judgment, visual discrimination, spatial-match, forward-span, instruction-following, and memory.
  Interventions: Behavioral: Physical Exercise Intervention; Behavioral: Cognitive Training Intervention
- Physical Exercise and Cognitive Control (Active Comparator): Physical Exercise Intervention: The physical exercise portion of the combined intervention consists of 45 minutes of multi-modal physical exercise focused on seated aerobic and progressive resistance training designed to improve aerobic capacity, muscular strength and endurance consistent with current exercise recommendations. The study team will deliver 3 sessions per week for 3 months.
  Cognitive Control: This consists of up to 20 minutes of puzzles and games, 2 days per week for 3 months. The participants will use on-line Brain HQ Control Games hosted by Posit Science, Inc. as an attention control.
  Interventions: Behavioral: Physical Exercise Intervention; Behavioral: Cognitive Control
- Cognitive Training and Stretching Control (Active Comparator): Stretching Control: This consists of up to 10 minutes of gentle stretching. The study team will deliver 3 sessions per week for 3 months.
  Cognitive Intervention: The cognitive portion of the combined intervention consists of a suite of 24 programs called Brain HQ developed by Posit Science Inc., organized into six categories: attention, speed, memory, people skills, intelligence, and navigation. The DDD-ECT trial will use 45-minute sessions of Brain HQ exercises. The modules are designed to improve time-order judgment, visual discrimination, spatial-match, forward-span, instruction-following, and memory. ly directing one session per week and available as needed for rest of the sessions.
  Interventions: Behavioral: Cognitive Training Intervention; Behavioral: Stretching Control
- Cognitive Control and Stretching Control (Sham Comparator): Stretching Control: This consists of up to 10 minutes of stretching. The study team will deliver 3 sessions per week for 3 months.
  Cognitive Control: This consists of up to 20 minutes of puzzles and games, 2 days per week for 3 months. The participants will use on-line Brain HQ Control Games hosted by Posit Science, Inc. as an attention control.
  Interventions: Behavioral: Stretching Control; Behavioral: Cognitive Control

INTERVENTIONS:
Behavioral: Physical Exercise Intervention — In home exercise intervention.
  Arms: Physical Exercise and Cognitive Control; Physical Exercise and Cognitive Training
Behavioral: Cognitive Training Intervention — Online cognitive training modules.
  Other Names: Brain HQ
  Arms: Cognitive Training and Stretching Control; Physical Exercise and Cognitive Training
Behavioral: Stretching Control — In home stretching.
  Arms: Cognitive Control and Stretching Control; Cognitive Training and Stretching Control
Behavioral: Cognitive Control — Online control puzzles and games.
  Other Names: Brain HQ
  Arms: Cognitive Control and Stretching Control; Physical Exercise and Cognitive Control

SUMMARY:
Primary Specific Aim: Determine the effect of the combined physical exercise and cognitive training on the cognitive function of ICU survivors aged 50 and older. Hypothesis: In comparison to older ICU survivors randomized to attention control or either intervention alone, those randomized to 12 weeks of combined physical exercise and cognitive training will have higher total index cognitive scores as assessed by the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) at 3 and 6 months post randomization.

Secondary Specific Aim 1: Determine the effect of the combined physical exercise and cognitive training on physical performance, anxiety and depressive symptoms, and quality of life of ICU survivors aged 50 and older. Hypotheses: In comparison to older ICU survivors randomized to attention control or either intervention alone, those randomized to 12 weeks of combined physical exercise and cognitive training will have higher physical performance as measured by short physical performance battery (SPPB) and two-minute step test, lower mood and anxiety symptoms as measured by Patient Health Questionnaire (PHQ-9) and Generalized Anxiety Disorder (GAD-7) scale, and higher quality of life as measured by the Medical Outcomes Study 36-item short form (SF-36) at 3 and 6-months post randomization.

Exploratory Aim 2: To examine the mechanisms of action of combined training. Hypothesis: At the completion of treatment, the combined intervention group will show reduced serum levels of CRP, IL-1, IL-6, IL-8, TNF-α, S-100β, and GFAP and increased levels of BDNF, VEGF, and IGF-1 compared to the attention control, or either intervention alone groups.

DETAILED DESCRIPTION:
Critical illness has deleterious consequences on both acute and chronic cognitive functions. Acute cognitive dysfunction manifests itself as delirium in the critically ill especially the elderly. Delirium is a complex neuropsychiatric syndrome characterized by acute and fluctuating changes in cognition and consciousness. 60% to 80% of critically ill ventilated older patients and 30% to 50% of those with less illness severity have delirium for at least one day of their ICU or hospital stay. Chronic cognitive dysfunction manifests as ICU acquired cognitive impairment and dementia after critical illness, affects multiple cognitive domains and persists years after hospital discharge. Up to 71% of critical illness survivors have cognitive impairment at one year after hospital discharge and close to 18% are diagnosed with new dementia including Alzheimer's disease within three years post ICU hospitalization.

Two million older Americans suffer from an episode of delirium during their intensive care unit (ICU) stay. Presence of delirium predisposes the elderly to immediate in-hospital complications including a longer length of ICU and hospital stay, increased risk of in-patient mortality and elevated costs of care. In addition, ICU delirium is associated with long-term post-discharge complications such as development of cognitive impairment and dementia. Current advances in the management of critical illness have notably improved the survival rates among this vulnerable segment of older adults. However, increased survival comes at a cost with as many as 70% of older ICU survivors who had an episode of delirium suffering from subsequent cognitive impairment and dementia. At present, there are no effective and scalable recovery models to remediate ICU acquired cognitive impairment and its attendant elevated dementia or Alzheimer's disease risk.

The inability to develop efficacious interventions to reduce ICU acquired cognitive impairment may stem from a limited understanding of the link between acute brain dysfunction (delirium) and chronic brain dysfunction (ICU acquired cognitive impairment, dementia or Alzheimer's disease). The investigators propose a recovery intervention guided by the pathophysiologic mechanisms implicated in producing critical illness delirium and elevated risk of cognitive impairment. The intervention targets inflammation, glial dysfunction and astrocyte activation along with restoration of neurotrophic factors while training function directly across multiple cognitive domains to reduce the burden of cognitive impairment among ICU survivors of delirium.

Over the past five years, Indiana University Center for Aging Research has developed a research infrastructure focused on delirium and delirium associated cognitive impairment, encompassing the ICU and post-ICU periods. This includes developing a bio-repository of serum delirium biomarkers, ICU based delirium trials, and post-ICU exercise and cognitive therapy recovery models. Building upon prior work and based on the pathophysiologic mechanisms mentioned above, the investigators now propose a novel home-based combined physical exercise and cognitive training program for older ICU survivors to improve cognitive impairment.

The study team is proposing a 2x2 factorial design randomized controlled trial (RCT) called "Decreasing Alzheimer's Disease and Related Dementias after Delirium-Exercise and Cognitive Training (DDD-ECT)" to evaluate the efficacy of 12 weeks of combined physical exercise and cognitive training on the primary outcome of cognitive function among older ICU survivors who experienced delirium or subsyndromal delirium during their ICU stay. The investigators propose to deliver these interventions via a facilitator-led, small group format using internet-enabled, multiparty-videoconference delivered directly into the participants' homes to achieve the study aims listed in the summary.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 50 years
* Admitted to medical and/or surgical ICUs at Methodist, University, or Eskenazi hospitals
* Discharged home or to sub-acute rehabilitation, long-term acute care, or skilled nursing facility
* Able to provide consent or has a legally authorized representative to provide consent
* Access to a telephone (study provides computer and broadband)
* Have at least one episode of subsyndromal delirium or delirium as determined by the Confusion Assessment Method for the ICU-7 (CAM-ICU).

Exclusion Criteria:

* Diagnosis of cancer with short life expectancy
* Current chemotherapy or radiation therapy (confirmed by electronic medical record)
* History of dementing illnesses and other neurodegenerative disease such as Alzheimer's disease, Parkinson disease, or vascular dementia (confirmed by EMR), or current prescription of anti-dementia medication, or ruled out by Functional Activities Questionnaire (FAQ) score defining dementia
* History of bipolar disorder or schizophrenia (confirmed by EMR)
* Current alcohol consumption > 5 drinks per day (self reported and/or confirmed by EMR)
* Vision < 20/80 via Snellen card or confirmed by EMR
* Low hearing or communicative ability (examiner rated) that would interfere with interventions and outcome assessments
* Have any active and untreated American College of Sports Medicine absolute contraindications to exercise (confirmed by EMR) including: acute myocardial infarctions within the past 2 days, ongoing unstable angina, uncontrolled cardiac arrhythmia with hemodynamic compromise, active endocarditis, symptomatic severe aortic stenosis, decompensated heart failure, acute pulmonary embolism, pulmonary infarction, or deep venous thrombosis, acute myocarditis or pericarditis, acute aortic dissection, physical disability that precludes safe and adequate testing, or are unable to obtain provider clearance for physical exercise for any contraindication where medical management is unclear
* Have any active and untreated American College of Sports Medicine relative contraindications to exercise (confirmed by EMR) including: known obstructive left main coronary stenosis, moderate to severe aortic stenosis with uncertain relationship to symptoms, tachydysrhythmias with uncontrolled ventricular rates, acquired advanced or complete heart block, recent stroke or transient ischemia attack, mental impairment with limited ability to cooperate, resting hypertension with systolic >200 mm Hg or diastolic >100 mm Hg, uncorrected medical conditions, such as significant anemia, important electrolyte imbalance, and hyperthyroidism, or are unable to obtain provider clearance for physical exercise for any contraindication where medical management is unclear
* Recovering from a skeletal fracture (confirmed by EMR), unless cleared by their physician of record to safely participate in exercise
* Acquired neurologic injury (stroke, traumatic brain injury, cerebral edema/swelling, anoxic brain injury, or any other acute/subacute severe neurologic deficit) as the admitting diagnosis or a new event during the course of hospitalization (confirmed by EMR)
* History of drug abuse within the last 3 months confirmed by EMR or self-report with Drug Abuse and Screening Test (DAST-10) score ≥ 3
* Have any spinal cord injury with persistent neurologic deficit at the time of study enrollment
* Status post tracheostomy and not eligible for a speaking valve
* Pregnant or nursing
* Incarcerated or homeless at time of study
* Lives outside the greater Indianapolis area

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Indiana University Health West Hospital, Avon, Indiana
  - Indiana University Health North Hospital, Carmel, Indiana
  - Indiana University Health Saxony Hospital, Fishers, Indiana
  - Eskenazi Health, Indianapolis, Indiana
  - Indiana University Health Methodist Hospital, Indianapolis, Indiana
  - Indiana University Health University Hospital, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khan SH, Perkins AJ, Unverzagt FW, Wang S, Moser LR, Moiz S, Jawaid S, Corlett D, Clark DO, Boustani MA, Gao S, Khan BA. Improving Recovery and Outcomes Every Day After the ICU (IMPROVE): A Randomized Controlled Trial. Crit Care Med. 2025 Aug 1;53(8):e1542-e1553. doi: 10.1097/CCM.0000000000006698. Epub 2025 May 22. PMID 40402024
- [Derived] Wang S, Hammes J, Khan S, Gao S, Harrawood A, Martinez S, Moser L, Perkins A, Unverzagt FW, Clark DO, Boustani M, Khan B. Improving Recovery and Outcomes Every Day after the ICU (IMPROVE): study protocol for a randomized controlled trial. Trials. 2018 Mar 27;19(1):196. doi: 10.1186/s13063-018-2569-8. PMID 29580264

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Per protocol subjects were considered to be enrolled in the study at the time of completion of the informed consent process. 249 subjects were enrolled. 153 subjects were randomized to one of the four study groups.
Groups:
- Physical Exercise and Cognitive Training: Physical Exercise Intervention: The physical exercise portion of the combined intervention consists of 45 minutes of multi-modal physical exercise focused on seated aerobic and progressive resistance training designed to improve aerobic capacity, muscular strength and endurance consistent with current exercise recommendations. The study team will deliver 3 sessions per week for 3 months.
  Cognitive Intervention: The cognitive portion of the combined intervention consists of a suite of 24 programs called Brain HQ developed by Posit Science Inc., organized into six categories: attention, speed, memory, people skills, intelligence, and navigation. The DDD-ECT trial will use 45-minute sessions of Brain HQ exercises. The modules are designed to improve time-order judgment, visual discrimination, spatial-match, forward-span, instruction-following, and memory.
  Physical Exercise Intervention: In home exercise intervention.
  Cognitive Training Intervention: Online cognitive training modules.
- Physical Exercise and Cognitive Control: Physical Exercise Intervention: The physical exercise portion of the combined intervention consists of 45 minutes of multi-modal physical exercise focused on seated aerobic and progressive resistance training designed to improve aerobic capacity, muscular strength and endurance consistent with current exercise recommendations. The study team will deliver 3 sessions per week for 3 months.
  Cognitive Control: This consists of up to 20 minutes of puzzles and games, 2 days per week for 3 months. The participants will use on-line Brain HQ Control Games hosted by Posit Science, Inc. as an attention control.
  Physical Exercise Intervention: In home exercise intervention.
  Cognitive Control: Online control puzzles and games.
- Cognitive Training and Stretching Control: Stretching Control: This consists of up to 10 minutes of gentle stretching. The study team will deliver 3 sessions per week for 3 months.
  Cognitive Intervention: The cognitive portion of the combined intervention consists of a suite of 24 programs called Brain HQ developed by Posit Science Inc., organized into six categories: attention, speed, memory, people skills, intelligence, and navigation. The DDD-ECT trial will use 45-minute sessions of Brain HQ exercises. The modules are designed to improve time-order judgment, visual discrimination, spatial-match, forward-span, instruction-following, and memory. ly directing one session per week and available as needed for rest of the sessions.
  Cognitive Training Intervention: Online cognitive training modules.
  Stretching Control: In home stretching.
- Cognitive Control and Stretching Control: Stretching Control: This consists of up to 10 minutes of stretching. The study team will deliver 3 sessions per week for 3 months.
  Cognitive Control: This consists of up to 20 minutes of puzzles and games, 2 days per week for 3 months. The participants will use on-line Brain HQ Control Games hosted by Posit Science, Inc. as an attention control.
  Stretching Control: In home stretching.
  Cognitive Control: Online control puzzles and games.
Period: Overall Study
Arm/Group | Physical Exercise and Cognitive Training | Physical Exercise and Cognitive Control | Cognitive Training and Stretching Control | Cognitive Control and Stretching Control
Started | 41 | 41 | 36 | 35
Completed | 28 | 30 | 27 | 24
Not Completed | 13 | 11 | 9 | 11
Not completed — missed | 1 | 2 | 0 | 1
Not completed — Lost to Follow-up | 2 | 2 | 1 | 0
Not completed — refusal | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 8 | 2 | 5 | 4
Not completed — Physician Decision | 1 | 2 | 2 | 2
Not completed — Death | 1 | 2 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Physical Exercise and Cognitive Training | Physical Exercise and Cognitive Control | Cognitive Training and Stretching Control | Cognitive Control and Stretching Control | Total
Number analyzed (Participants) | 41 | 41 | 36 | 35 | 153
Age, Continuous [Mean (Full Range); unit: years] | 64.3 [50 to 83] | 64.4 [50 to 83] | 64.6 [50 to 89] | 65.4 [52 to 81] | 64.7 [50 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 29 | 22 | 18 | 100
  Male | 10 | 12 | 14 | 17 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 41 | 41 | 36 | 35 | 153
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 10 | 14 | 13 | 17 | 54
  White | 30 | 27 | 21 | 17 | 95
  More than one race | 1 | 0 | 2 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 41 | 41 | 36 | 35 | 153

OUTCOME MEASURES:

1. Primary Outcome: Cognitive Status Outcome at 6 Months
Description: The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) will measure cognitive status.
  The z-scores for the subscales have a mean of 0 and standard deviation of 1. The overall z-score is the mean of the 7-item z-scores. Z-scores above the standard deviation represent better cognitive outcomes.
Time Frame: 6 months post study randomization
Population: Only participants who were able to complete the scale are included in the analysis.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Physical Exercise and Cognitive Training | Physical Exercise and Cognitive Control | Cognitive Training and Stretching Control | Cognitive Control and Stretching Control
Number analyzed (Participants) | 27 | 30 | 27 | 24
Z-score | 0.24 (0.64) | 0.36 (0.59) | 0.21 (0.58) | 0.35 (0.64)
Statistical Analysis 1: Comparison: Physical Exercise and Cognitive Training vs Physical Exercise and Cognitive Control vs Cognitive Training and Stretching Control vs Cognitive Control and Stretching Control; Test type: Superiority; p = 0.747, Mixed Models Analysis

2. Primary Outcome: Cognitive Status Outcome at 3 Months
Description: as for outcome 1
Time Frame: 3 months post study randomization
Population: Only participants who were able to complete the scale are included in the analysis.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Physical Exercise and Cognitive Training | Physical Exercise and Cognitive Control | Cognitive Training and Stretching Control | Cognitive Control and Stretching Control
Number analyzed (Participants) | 27 | 28 | 27 | 25
Z-score | -0.21 (0.69) | 0.28 (0.58) | -0.13 (0.65) | -0.07 (0.59)
Statistical Analysis 1: Comparison: Physical Exercise and Cognitive Training vs Physical Exercise and Cognitive Control vs Cognitive Training and Stretching Control vs Cognitive Control and Stretching Control; Test type: Superiority; p = 0.032, Mixed Models Analysis

3. Secondary Outcome: Physical Performance Scores at 3 Months
Description: The Short Physical Performance Battery (SPPB) will measure physical training effects on balance and strength.
  Ranges from 0-12: higher score is better outcome
Time Frame: 3 month post study randomization
Population: Only participants who were able to complete the scale are included in the analysis. Post COVID-19 no SPPB or 2 Minute Step Tests were performed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Exercise and Cognitive Training | Physical Exercise and Cognitive Control | Cognitive Training and Stretching Control | Cognitive Control and Stretching Control
Number analyzed (Participants) | 10 | 15 | 12 | 11
score on a scale | 6.60 (4.86) | 7.80 (4.18) | 4.92 (4.46) | 8.18 (3.37)
Statistical Analysis 1: Comparison: Physical Exercise and Cognitive Training vs Physical Exercise and Cognitive Control vs Cognitive Training and Stretching Control vs Cognitive Control and Stretching Control; Test type: Superiority; p = 0.264, Mixed Models Analysis

4. Secondary Outcome: Physical Performance Scores at 6 Months
Description: as for outcome 3
Time Frame: 6 month post study randomization
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Exercise and Cognitive Training | Physical Exercise and Cognitive Control | Cognitive Training and Stretching Control | Cognitive Control and Stretching Control
Number analyzed (Participants) | 12 | 14 | 7 | 12
score on a scale | 5.00 (4.99) | 7.07 (4.53) | 6.57 (3.31) | 7.00 (4.31)
Statistical Analysis 1: Comparison: Physical Exercise and Cognitive Training vs Physical Exercise and Cognitive Control vs Cognitive Training and Stretching Control vs Cognitive Control and Stretching Control; Test type: Superiority; p = 0.511, Mixed Models Analysis

5. Secondary Outcome: Cardiovascular Fitness Scores at 3 Months
Description: The 2-Minute Step Test will measure physical training effects on cardiovascular fitness.
  Number of steps, higher = better outcome
Time Frame: 3 month post study randomization
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: number of steps in place in 2 minutes
Arm/Group | Physical Exercise and Cognitive Training | Physical Exercise and Cognitive Control | Cognitive Training and Stretching Control | Cognitive Control and Stretching Control
Number analyzed (Participants) | 10 | 12 | 12 | 9
number of steps in place in 2 minutes | 47.30 (38.27) | 45.67 (43.08) | 27.67 (38.00) | 41.44 (27.75)
Statistical Analysis 1: Comparison: Physical Exercise and Cognitive Training vs Physical Exercise and Cognitive Control vs Cognitive Training and Stretching Control vs Cognitive Control and Stretching Control; Test type: Superiority; p = 0.677, Mixed Models Analysis

6. Secondary Outcome: Cardiovascular Fitness Scores at 6 Months
Description: as for outcome 5
Time Frame: 6 month post study randomization
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: number of steps in place in 2 minutes
Arm/Group | Physical Exercise and Cognitive Training | Physical Exercise and Cognitive Control | Cognitive Training and Stretching Control | Cognitive Control and Stretching Control
Number analyzed (Participants) | 12 | 13 | 7 | 11
number of steps in place in 2 minutes | 35.25 (36.86) | 40.00 (37.21) | 36.29 (31.28) | 32.36 (39.16)
Statistical Analysis 1: Comparison: Physical Exercise and Cognitive Training vs Physical Exercise and Cognitive Control vs Cognitive Training and Stretching Control vs Cognitive Control and Stretching Control; Test type: Superiority; p = 0.815, Mixed Models Analysis

7. Secondary Outcome: Depression Scores at 3 Months
Description: The Patient Health Questionnaire-9 (PHQ-9) will measure intervention effects on depression levels.
  Ranges from 0-27, higher score is worse outcome
Time Frame: 3 month post study randomization
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Exercise and Cognitive Training | Physical Exercise and Cognitive Control | Cognitive Training and Stretching Control | Cognitive Control and Stretching Control
Number analyzed (Participants) | 27 | 29 | 28 | 25
score on a scale | 7.19 (6.73) | 6.03 (4.91) | 5.36 (4.98) | 5.84 (5.01)
Statistical Analysis 1: Comparison: Physical Exercise and Cognitive Training vs Physical Exercise and Cognitive Control vs Cognitive Training and Stretching Control vs Cognitive Control and Stretching Control; Test type: Superiority; p = 0.719, Mixed Models Analysis

8. Secondary Outcome: Depression Scores at 6 Months
Description: as for outcome 7
Time Frame: 6 month post study randomization
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Exercise and Cognitive Training | Physical Exercise and Cognitive Control | Cognitive Training and Stretching Control | Cognitive Control and Stretching Control
Number analyzed (Participants) | 28 | 30 | 27 | 24
score on a scale | 7.79 (6.06) | 5.90 (4.93) | 5.04 (6.45) | 5.67 (5.58)
Statistical Analysis 1: Comparison: Physical Exercise and Cognitive Training vs Physical Exercise and Cognitive Control vs Cognitive Training and Stretching Control vs Cognitive Control and Stretching Control; Test type: Superiority; p = 0.346, Mixed Models Analysis

9. Secondary Outcome: Anxiety Scores at 3 Months
Description: The Generalized Anxiety Disorder Scale (GAD-7) will measure intervention effects on anxiety levels.
  Ranges from 0-21, higher score is worse outcome
Time Frame: 3 month post study randomization
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Exercise and Cognitive Training | Physical Exercise and Cognitive Control | Cognitive Training and Stretching Control | Cognitive Control and Stretching Control
Number analyzed (Participants) | 27 | 29 | 28 | 25
score on a scale | 4.27 (5.39) | 4.48 (5.91) | 3.32 (4.37) | 4.24 (4.82)
Statistical Analysis 1: Comparison: Physical Exercise and Cognitive Training vs Physical Exercise and Cognitive Control vs Cognitive Training and Stretching Control vs Cognitive Control and Stretching Control; Test type: Superiority; p = 0.910, Mixed Models Analysis

10. Secondary Outcome: Anxiety Scores at 6 Months
Description: as for outcome 9
Time Frame: 6 month post study randomization
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Exercise and Cognitive Training | Physical Exercise and Cognitive Control | Cognitive Training and Stretching Control | Cognitive Control and Stretching Control
Number analyzed (Participants) | 28 | 30 | 27 | 24
score on a scale | 4.25 (5.64) | 4.33 (5.41) | 3.48 (5.91) | 3.13 (4.20)
Statistical Analysis 1: Comparison: Physical Exercise and Cognitive Training vs Physical Exercise and Cognitive Control vs Cognitive Training and Stretching Control vs Cognitive Control and Stretching Control; Test type: Superiority; p = 0.794, Mixed Models Analysis

11. Secondary Outcome: Quality of Life Scores at 3 Months
Description: The Medical Outcomes Study 36 item short form (SF-36) will measure participant quality of life scores.
  range of 0 - 100 (higher = better outcome)
Time Frame: 3 month post study randomization
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Exercise and Cognitive Training | Physical Exercise and Cognitive Control | Cognitive Training and Stretching Control | Cognitive Control and Stretching Control
Number analyzed (Participants) | 27 | 29 | 28 | 25
score on a scale | 34.49 (12.51) | 34.25 (12.37) | 31.74 (11.42) | 33.57 (11.49)
Statistical Analysis 1: Comparison: Physical Exercise and Cognitive Training vs Physical Exercise and Cognitive Control vs Cognitive Training and Stretching Control vs Cognitive Control and Stretching Control; Test type: Superiority; p = 0.626, Mixed Models Analysis

12. Secondary Outcome: Quality of Life Scores at 6 Months
Description: as for outcome 11
Time Frame: 6 month post study randomization
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Exercise and Cognitive Training | Physical Exercise and Cognitive Control | Cognitive Training and Stretching Control | Cognitive Control and Stretching Control
Number analyzed (Participants) | 28 | 30 | 27 | 23
score on a scale | 34.72 (13.14) | 34.08 (11.64) | 33.36 (10.77) | 34.40 (9.97)
Statistical Analysis 1: Comparison: Physical Exercise and Cognitive Training vs Physical Exercise and Cognitive Control vs Cognitive Training and Stretching Control vs Cognitive Control and Stretching Control; Test type: Superiority; p = 0.774, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Participants were assessed for adverse events from the time of informed consent process completion until the end of study participation. This was approximately 6 months if the study was completed.
Arm/Group | Physical Exercise and Cognitive Training | Physical Exercise and Cognitive Control | Cognitive Training and Stretching Control | Cognitive Control and Stretching Control
All-Cause Mortality (participants affected / at risk) | 1/41 | 2/41 | 1/36 | 3/35
Serious Adverse Events (participants affected / at risk) | 0/41 | 1/41 | 0/36 | 0/35
Other Adverse Events (participants affected / at risk) | 2/41 | 3/41 | 1/36 | 0/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Physical Exercise and Cognitive Training (N=41) | Physical Exercise and Cognitive Control (N=41) | Cognitive Training and Stretching Control (N=36) | Cognitive Control and Stretching Control (N=35)
elevated heart rate (Cardiac disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Physical Exercise and Cognitive Training (N=41) | Physical Exercise and Cognitive Control (N=41) | Cognitive Training and Stretching Control (N=36) | Cognitive Control and Stretching Control (N=35)
elevated heart rate (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
O2 saturation lower than 88% (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-12-01): https://cdn.clinicaltrials.gov/large-docs/17/NCT03095417/Prot_SAP_001.pdf
  • Informed Consent Form (2019-01-30): https://cdn.clinicaltrials.gov/large-docs/17/NCT03095417/ICF_000.pdf